CLINICAL TRIAL: NCT00785070
Title: Pre and Post Orthopedic Surgery Sleep and Cardiac Testing (PROSPECT)
Acronym: PROSPECT
Status: Completed | Type: Observational
Sponsor: Memorial Health System (Other)
Collaborators: Nexan Inc (Industry)
Responsible Party: C. Bryan Carr, M.D., Memorial Health System
Other Study IDs: PROSPECT
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2009-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: Perioperative; Obstructive Sleep Apnea; Screening; Home Sleep Testing
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Perioperative

SUMMARY:
* Evaluate sleep disordered breathing before and after orthopedic surgery utilizing a FDA cleared to market (510k) home sleep study device (Nexan Inc., ClearPath System)
* Compare Berlin Questionnaire and Epworth Sleep Scale questionnaires to the home sleep study device results.
* Evaluate effectiveness of the home sleep study testing in the orthopedic presurgical population.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing knee or hip total joint replacement
* Answer Yes to any PROSPECT health history questions and/or score Positive on the sleep questionnaires

Exclusion Criteria:

* Tape Allergy
* Previous Diagnosis Of Obstructive Sleep Apnea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Orthopedic Total Hip or Knee Joint Replacement
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Comparison of objective sleep data to standardized sleep questionnaires | Pre and Post Operative

SECONDARY OUTCOMES:
Compare Pre and Post Operative Objective sleep data | Pre and post operative

CONTACTS AND LOCATIONS:
Overall Officials: Clayton B. Carr, M.D., Principal Investigator — Memorial Health System
Locations (1):
- Memorial Health System, Colorado Springs, Colorado, United States